CLINICAL TRIAL: NCT03260829
Title: Evaluation of the Effect of Local Injected Vitamin C on Accelerating the Orthodontic Movement of Maxillary Canine Impaction: A Clinical Trial
Brief Title: Efficacy of Injectable Vitamin C on Accelerating Canine Movement: A Clinical Study
Acronym: mesotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, nermin mohammed ahmed yussif, assistant lecturer, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: oral and dental medicine; no conflict of interest (Other)
Record Dates: First submitted 2017-01-11; First posted 2017-08-24 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Palatally Impacted Canines
Keywords: vitamin C; palatally impacted canines; intraepidermal injection
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin C injection (Active Comparator): orthodontic traction with vitamin C injection
  Interventions: Drug: vitamin C
- orthodontic traction (Placebo Comparator): orthodontic traction without vitamin C injection
  Interventions: Drug: vitamin C

INTERVENTIONS:
Drug: vitamin C — 25 IU of vitamin C injected intraepidermally for 6-8 visits till eruption achieved
  Other Names: ascorbic acid

SUMMARY:
efficacy of the injectable vitamin C to reduce the time of canine traction

DETAILED DESCRIPTION:
Objective. The purpose of this study is to investigate the role and efficiency of the locally injected vitamin C in the enhancement of the palatally impacted canine movement.

Design. Twelve adult patients with unilateral palatally impacted canines were included in this study. The enrolled patients were randomly allocated into the study groups; control group; orthodontic traction and he test group: orthodontic traction enhanced by intraepidermic vitamin C injection. The study duration was 12 months.

ELIGIBILITY:
Inclusion Criteria:

* medically free
* patient with good to fair oral hygiene (gingivitis may be included)
* both sexes were included
* unilateral palatally positioned permenant canines
* absence of previous orthodontic treatment
* absence of supernumerary teeth, odontoms, cysts, traumatic injuries
* the α angle within grade II to III

Exclusion Criteria:

* systemic diseases especially diabetes and bone diseases
* pregnant and lactating mothers
* Local causes (smoking, mouth breathing, local trauma and periodontitis).

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
rate of tooth movement | 12 months
  the achieved movement in millimeters in one year

SECONDARY OUTCOMES:
level of alveolar bone | 12 months
  the level of the interproximal and facial alveolar bone after orthodontic treatment with or without injection

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine, Giza, Giza Governorate, Egypt

REFERENCES:
- [Result] Makar AB, McMartin KE, Palese M, Tephly TR. Formate assay in body fluids: application in methanol poisoning. Biochem Med. 1975 Jun;13(2):117-26. doi: 10.1016/0006-2944(75)90147-7. No abstract available.